CLINICAL TRIAL: NCT05998720
Title: Application of New Magnetic Resonance Technique-UTE in Hip Joint Lesions
Brief Title: Application of New Magnetic Resonance UTE Technique in Hip Joint Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.FSK.025
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Hip Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal group: There are no lesions on the hip.
- abnormal group: There are some lesions on the hip.

SUMMARY:
Explore the imaging and quantitative monitoring of hip bone, cartilage and ligament by magnetic resonance UTE technology, combined with QCT and DXA technology, to provide a more accurate basis for clinical evaluation and treatment.

DETAILED DESCRIPTION:
Osteoporosis is a systemic bone metabolism-related disease characterized by decreased bone mass per unit volume, increased bone fragility, decreased bone density, thinning of the bone cortex and changes in bone microstructure. It often occurs in the lumbar spine and hip joint. Femoral neck fracture is a common complication of hip osteoporosis, which seriously affects people's quality of life. UTE technology can clearly image and quantify human cortical bone and cancellous bone, and advanced UTE technology such as STAIR-UTE and UTE-MT have made some progress in the field of osteoporosis. The purpose of this study was to explore UTE technology for imaging and quantitative study of cortical bone, cancellous bone and cartilage of hip joint, and to find more accurate imaging methods for clinical evaluation of hip osteoporosis and other diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with past or suspected osteoporosis and bone loss;
2. Patients with previous femoral neck fracture;
3. Patients with avascular necrosis of femoral head;
4. Hip osteoarthritis patients.

Exclusion Criteria:

1. Patients with metal implants in corresponding parts;
2. Claustrophobic.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2024-06-13 (Estimated)

PRIMARY OUTCOMES:
proton density fat fraction (PDFF) | Baseline (before surgery)
  Magnetic resonance proton density fat fraction
T2 relaxation rate | Baseline (before surgery)
  R2*
Magnetization Transfer Ratio (MTR) | Baseline (before surgery)
  magnetization transfer ratio
T1rho | Baseline (before surgery)
  spin-lattice relaxation in the rotation ame

SECONDARY OUTCOMES:
Subjective rating values | Baseline (before surgery)
  rating values

CONTACTS AND LOCATIONS:
Overall Officials: Shaolin Li, Study Director — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Radiography department, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No